CLINICAL TRIAL: NCT00585091
Title: The Development of Tolerance to α1-Adrenoceptor Blockade With Chronic Carvedilol Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, edward gilbert, Professor of Medicine, University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00011909; IRB# 00011909
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Other): All patients undergo repeated phenylephrine infusions during standard up-titration and maintenance of carvedilol treatment.
  Interventions: Drug: phenylephrine

INTERVENTIONS:
Drug: phenylephrine — All patients undergo repeated phenylephrine infusions during standard up-titration and maintenance of carvedilol treatment.

SUMMARY:
There is now strong evidence from clinical trials that carvedilol therapy in heart failure is superior to therapy with metoprolol. Not only does carvedilol have superior effects on lipid profiles, insulin sensitivity, renal blood flow, and reversal of pathologic remodeling but also its use is associated with fewer deaths compared to metoprolol. These facts make it important to carefully define how metoprolol and carvedilol are pharmacologically different. One potential difference is α1-AR antagonism. If we demonstrate that these α1-AR effects are preserved with chronic therapy, then α1-AR blockade may have an important role in carvedilol favorably altering the natural history of heart failure. On the other hand, if we demonstrate that tolerance to the α1-AR blockade effect of carvedilol decreases with time, then it would be unlikely that this pharmacologic property contributes to the efficacy of carvedilol. In such a case other pharmacologic properties, such as antioxidant activity, would appear to be important. These results will help guide future studies into CHF and AR blockade.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 85 years
2. Symptomatic heart failure, NYHA class I to III
3. Left ventricular ejection fraction < 0.40
4. Give written informed consent

Exclusion Criteria:

1. active myocarditis
2. congenital heart disease
3. uncorrected, hemodynamically significant stenotic valvular disease
4. hypertrophic cardiomyopathy
5. Asthma or other obstructive airway diseases requiring bronchodilators
6. Heart rate < 60 beats/min, supine systolic blood pressure < 85 mm Hg, supine diastolic blood pressure > 90 mm Hg
7. Uncontrolled Hypertension (Systolic BP >140 mmHg, Diastolic BP > 90 mmHg).
8. Sick sinus syndrome, Mobitz type 2 second degree AV block or third degree AV block unless controlled with an artificial implantable pacemaker
9. NYHA functional class IV symptoms
10. Treatment with an excluded medication (see Excluded Medications below)
11. Myocardial infarction or coronary artery intervention (CABG or angioplasty) within three months
12. Unstable angina pectoris
13. Presence of any progressive systemic disease that would be expected to impact the patient's outcome over the time course of the study
14. Uncorrected endocrine disorders including primary aldosteronism, pheochromocytoma, hyperthyroidism, hypothyroidism, brittle type 1 diabetes mellitus
15. Evidence of significant renal disease (serum creatinine > 2.5 mg/dl), or hepatic disease (transaminase level > three fold higher than laboratory normal)
16. Symptomatic peripheral vascular disease
17. Inability or unwillingness to cooperate with study or give written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-10; Primary Completion 2007-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine if tolerance to α1-AR blockade develops with the chronic administration of carvedilol in heart failure patients. | Oct 2003-Aug 2008

SECONDARY OUTCOMES:
All patients undergo repeated phenylephrine infusions during standard up-titration and maintenance of carvedilol treatment. | Oct 2003-Aug 2008

CONTACTS AND LOCATIONS:
Overall Officials: Mark Munger, PharmD, Principal Investigator — Professor, Pharmacotherapy
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Van Tassell BW, Rondina MT, Huggins F, Gilbert EM, Munger MA. Carvedilol increases blood pressure response to phenylephrine infusion in heart failure subjects with systolic dysfunction: evidence of improved vascular alpha1-adrenoreceptor signal transduction. Am Heart J. 2008 Aug;156(2):315-21. doi: 10.1016/j.ahj.2008.04.004. Epub 2008 Jun 20. PMID 18657662